CLINICAL TRIAL: NCT00000376
Title: Cognitive and Drug Therapy for Drug-Resistant Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R21MH052737 (NIH); R21MH052737 (NIH); DSIR
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2005-12

CONDITIONS: Depression; Anxiety Disorders; Personality Disorders; Drug-resistant Depression
Keywords: Adult; Antidepressive Agents, Tricyclic; Anxiety Disorders; Cognitive Therapy; Combined Modality Therapy; Depression; Desipramine; Female; Human; Male; Personality Disorders; Pilot Projects; Patient Care Team; Antidepressive Agents, Tricyclic -- *therapeutic use; Depression -- *therapy; Depression -- drug therapy; Desipramine -- *therapeutic use
MeSH Terms: conditions — Depression; Anxiety Disorders; Personality Disorders | interventions — Cognitive Behavioral Therapy; Desipramine

INTERVENTIONS:
Behavioral: Cognitive therapy
Drug: Desipramine

SUMMARY:
To develop an effective combined cognitive therapy (CT) plus drug treatment for patients with drug-resistant depression (DRD) (i.e., depression that is refractory to medication). To develop a manual for combined treatment for DRD that integrates three existing forms of CT (CT for depression, CT for personality disorders, and CT for anxiety disorders), and that specifies interventions for combining CT and medication when two therapists (psychotherapist and pharmacotherapist) provide the treatment. To obtain outpatient, randomized control, pilot data on the clinical value of the combined CT plus drug treatment, using the standard antidepressant desipramine (DMI), to obtain effect sizes and to determine if the treatment merits further investigation in a clinical trial. To develop a therapist adherence measure for the combined treatment.

Patients receive 1 of 2 treatments: CT plus DMI (n = 18) or DMI plus Clinical Management (n = 12). The first 6 of the 18 CT plus DMI patients are treated in a pre-pilot phase before randomization begins. All treatments continue for 6 months. The major assessment battery is administered at intake, 3 months, 6 months, and follow-up 6 months later. All treatments are closely monitored via audiotapes and supervision for purposes of developing and refining the CT plus drug treatment. The audiotapes are also used for development of the adherence measure. The primary outcome measures are Hamilton Rating Scale for Depression scores, Beck Depression Inventory scores, percent of patients who achieve clinical remission of symptoms, and percent showing attrition from treatment. Compliance with the treatment regimens is also a targeted and measured outcome variable.

DETAILED DESCRIPTION:
To develop an effective combined cognitive therapy (CT) plus drug treatment for patients with drug-resistant depression (DRD) (i.e., depression that is refractory to medication). To develop a manual for combined treatment for DRD that integrates three existing forms of CT (CT for depression, CT for personality disorders, and CT for anxiety disorders), and that specifies interventions for combining CT and medication when two therapists (psychotherapist and pharmacotherapist) provide the treatment. To obtain outpatient, randomized control, pilot data on the clinical value of the combined CT plus drug treatment, using the standard antidepressant desipramine (DMI), to obtain effect sizes and to determine if the treatment merits further investigation in a clinical trial. To develop a therapist adherence measure for the combined treatment.

Patients receive 1 of 2 treatments: CT plus DMI (n = 18) or DMI plus Clinical Management (n = 12). The first 6 of the 18 CT plus DMI patients are treated in a pre-pilot phase before randomization begins. All treatments continue for 6 months. The major assessment battery is administered at intake, 3 months, 6 months, and follow-up 6 months later. All treatments are closely monitored via audiotapes and supervision for purposes of developing and refining the CT plus drug treatment. The audiotapes are also used for development of the adherence measure. The primary outcome measures are Hamilton Rating Scale for Depression scores, Beck Depression Inventory scores, percent of patients who achieve clinical remission of symptoms, and percent showing attrition from treatment. Compliance with the treatment regimens is also a targeted and measured outcome variable.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must have:

Drug-resistant depression (DRD).

Ages: 21 Years to 60 Years | Sex: All
Age Groups: Adult
Dates: Start 1996-03; Study Completion 1999-02

CONTACTS AND LOCATIONS:
Overall Officials: Karla Moras, PhD, Principal Investigator